CLINICAL TRIAL: NCT04864093
Title: Predicative Valute of Muscular Ultrasound in the Diagnosta of ICUAW in Critically Ill Patients
Brief Title: Muscular Ultrasound and Production of ICUAW
Acronym: MUICUAW
Status: Completed | Type: Observational
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Davide Chiumello, PROFESSOR, University of Milan
Other Study IDs: Umilan@
Record Dates: First submitted 2021-04-22; First posted 2021-04-28 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Weakness, Muscle
MeSH Terms: conditions — Muscle Weakness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: muscular ultrasound — respiratroy and muscular ultrasound

SUMMARY:
Skeletal muscle weakness is a common complication of acute respiratory failure, shock and other manifestations of critical illness or injury. ICU acquired weakness (ICUAW) - an entity defined as a bundle of critically illness neuro-myopathy and disuse atrophy - is generally diagnosed on the basis of a volitional, clinical strength evaluation, which however requires patient cooperation and ability to comprehend the assessor's instructions. As patients are often unconscious or uncooperative, due to sedation or delirium, such clinical diagnosis is often not possible or is delayed. A further subclassification of critical illness neuromyopathy can be achieved using detailed nonvolitional electrophysiological investigations, which can be challenging in the ICU as they require skilled personnel for both assessment and interpretation. An average Medical Research Council strength score (MRC-SS) combined for 12 specified muscle groups lower than 48 has been widely used for diagnosing ICUAW. Recent studies reported the clinical applicability of the MRC-SS in a general ICU population, in particular its clinical usefulness in predicting ICU and in-hospital patient outcomes . Moreover, interobserver agreement and clinical predictive value have already been showed (8). However, ICU general population is less likely to be able to cooperate with volitional strength assessment and more likely to have limited access to their extremities because of trauma, burns and treatment involving medical devices. For these reasons, MRC-SS may be confined to the later stages of ICU stay. Skeletal muscle ultrasound is used for the evaluation of muscular, tendon and joint disorders. It allows the evaluation of normal and pathological skeletal muscles through the measure of parameters reflecting size, such as cross sectional area (CSA) , and architecture by calculating the pennation angle, and it allows quick and repeated bedside evaluations. Despite such promising features, to date, there are few published studies that have reported the clinical applicability of the muscle ultrasound in prediction of ICUAW during the ICU stay. The principal aim of this study is to evaluate the variation of peripheral muscle ultrasound characteristics (such as CSA and pennation angle) during the ICU stay and its possible early predictive value of ICUAW as compared to the MRC-SS performed when patients are able to cooperate.

DETAILED DESCRIPTION:
Skeletal muscle weakness is a common complication of acute respiratory failure, shock and other manifestations of critical illness or injury. ICU acquired weakness (ICUAW) - an entity defined as a bundle of critically illness neuro-myopathy and disuse atrophy - is generally diagnosed on the basis of a volitional, clinical strength evaluation, which however requires patient cooperation and ability to comprehend the assessor's instructions. As patients are often unconscious or uncooperative, due to sedation or delirium, such clinical diagnosis is often not possible or is delayed. A further subclassification of critical illness neuromyopathy can be achieved using detailed nonvolitional electrophysiological investigations, which can be challenging in the ICU as they require skilled personnel for both assessment and interpretation. An average Medical Research Council strength score (MRC-SS) combined for 12 specified muscle groups lower than 48 has been widely used for diagnosing ICUAW. Recent studies reported the clinical applicability of the MRC-SS in a general ICU population, in particular its clinical usefulness in predicting ICU and in-hospital patient outcomes . Moreover, interobserver agreement and clinical predictive value have already been showed (8). However, ICU general population is less likely to be able to cooperate with volitional strength assessment and more likely to have limited access to their extremities because of trauma, burns and treatment involving medical devices. For these reasons, MRC-SS may be confined to the later stages of ICU stay. Skeletal muscle ultrasound is used for the evaluation of muscular, tendon and joint disorders. It allows the evaluation of normal and pathological skeletal muscles through the measure of parameters reflecting size, such as cross sectional area (CSA) , and architecture by calculating the pennation angle, and it allows quick and repeated bedside evaluations. Despite such promising features, to date, there are few published studies that have reported the clinical applicability of the muscle ultrasound in prediction of ICUAW during the ICU stay. The principal aim of this study is to evaluate the variation of peripheral muscle ultrasound characteristics (such as CSA and pennation angle) during the ICU stay and its possible early predictive value of ICUAW as compared to the MRC-SS performed when patients are able to cooperate.

Materials and methods

Study design and ethical approval

observational, single-center study in a mixed medical and surgical ICU in a university teaching hospital. We will investigate the variation of CSA and pennation angle of rectus femoris over the ICU stay. Moreover, we will examine the clinical predictive value of these two variables as compared with MRC-SS at awakening. Patients 18 years of age and older who had been invasively ventilated for 48 hours were eligible for inclusion. Exclusion criteria included preexisting neurological weakness, pregnancy, malignancy, and those admitted for routine overnight postoperative surgical recovery. A flow diagram of the study is showed in figure 1.

Study protocol

At ICU admission (T1), patients underwent muscular ultrasound comprehensive of rectus femoris cross sectional area (RFCSA) and pennation angle, diaphragm, and parasternal intercostal end-expiratory thickness appraisal. At the same time, anthropometric data and biochemical parameters necessary for the calculations of severity score (Sequential organ failure assessment -SOFA (16); Simplified acute physiology score- SAPS II ; Acute Physiology and Chronic Health Evaluation - APACHE II ) were collected. All the same measures were repeated at day 3 (T3) and 7 (T7).

Anthropometric Assessment

Anthropometric measurements of body length and weight will be recorded at ICU admission. The actual body weight as reported by the patients when able to do it was collected. From anthropometric data, body mass index (BMI, kg/m2) will be calculated, while ideal body weight was calculated using a standard formula as previously described .

Muscular ultrasound

RFCSA will bemeasured by B-mode ultrasonography using an 8 MHz, 5.6 cm linear transducer array (MindRay TE-5 machine, Mindray Bio-Medical Electronics Co. Ltd. Shenzen, China), similar to the method described elsewhere (11). The pennation angle, the angle of insertion of muscle fascicles into the deep aponeurosis, of the rectus femoris will be measure on the longitudinal view by rotating the probe parallel to either the lateral or medial head of the muscle on the position where we measured CSA. To obtain precise measurements of muscle parameters, all measurements will be performed by the same sonographer (PF) with 5 years of experience . All data will be measure three times, and the average value will be used for further analysis.

Diaphragm end-expiratory thickness will be measure in the right hemi-diaphragm in the zone of apposition as described elsewhere . All ultrasound examinations will be performe using a 10-15 MHz linear transducer in B mode (MindRay TE-5 machine, Mindray Bio-Medical Electronics Co. Ltd. Shenzen, China) by the same trained operators (PF). The inferior border of the costophrenic sinus will be identifiy as the zone of transition from the artefactual representation of the lung to the visualization of diaphragm and liver. The expiratory thickening of the parasternal intercostal muscles will be assesse with a linear probe placed 3 cm laterally from the sternum, and oriented along the sagittal plane, between the 2nd and the 3rd ribs (22). Muscle thickness will be measure just above the pleural line between the inner and outermost hyperechogenic layers of the muscle fascial borders. Images will be recorde for a subsequent computer-assisted quantitative analysis performed by a trained investigator (MU), unaware of the ventilatory condition.

MRC-SS

The consciousness level of patients will be determine using the Richmond Agitation Sedation Scale, with a score from -1 to +1 being indicative of wakefulness. Awake patients will then required to demonstrate a positive response to simple one-stage commands. Successful completion of commands was followed by muscle strength assessment using the MRC-SS - a six-point grading scale ranging from 0 (no visible contraction) to 5 (normal power) applied to six upper- and lower-limb muscle groups bilaterally (25). The day upon which MRC-SS will be performe will be recorded. ICUAW is defined as an MRC-SS less than 48 out of a possible score of 60. A standardized protocol for performing the MRC-SS will be always followed during testing. Given the volitional nature of manual muscle testing, strong verbal encouragement will be provided during all strength assessments.

statistical analysis

The computation of the study power isbased on the primary outcome (prediction of ICU-acquired weakness). A previous study found a correlation between diaphragm ultrasound and the development of ICU-acquired weakness of r=0.3. Since the current study also assesses peripheral muscle ultrasound, we hypothesized that a stronger correlation (about twice that found in the cited study) could be found with 80% power at a 5% significance level by enrolling 47 patients.

Data will be analyzed using Stata/SE 12.0 (StataCorp, College Station, TX USA) statistical software package. Two-tailed P-values <0.05 will be considered statistically significant. Normality will be assessed by the Shapiro-Francia test. Results will be reported as mean ± standard deviation if normally distributed, or median [25-75th percentiles] otherwise, and differences will be tested with a two-sided t test or the MannWhitney U test. Categorical variables are expressed as counts and percentage and the Chi-square or Fischer exact test will be used for analysis.

ELIGIBILITY:
Inclusion Criteria:

patients admitted to ICU witha prediction of ICU stay >7 days

Exclusion Criteria:

Exclusion criteria included preexisting neurological weakness, pregnancy, malignancy, and those admitted for routine overnight postoperative surgical recover

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all ICU patients
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2021-01-21 (Actual); Primary Completion 2021-10-21 (Actual); Study Completion 2021-10-21 (Actual)

PRIMARY OUTCOMES:
muscular reduction over the time | One year
  Muscular ultrasound detect a muscles reduction over the time

SECONDARY OUTCOMES:
muscular ultrasond predictivity of ICUAW | One year
  Muscular ultrasound evauation anticipate the diagnosta of ICUAW

CONTACTS AND LOCATIONS:
Locations (1):
- ASST Santi Paolo carlo, Milan, Italy

IPD SHARING:
Plan to Share IPD: No